CLINICAL TRIAL: NCT00933790
Title: A Randomized Controlled Clinical Trial Comparing Daily Vs. Intermittent 6 - Month Short Course Chemotherapy in Reducing Failures & Emergence of Acquired Rifampicin Resistance (ARR) in Patients With HIV and Pulmonary Tuberculosis
Brief Title: Comparing Daily vs Intermittent Regimen of ATT in HIV With Pulmonary Tuberculosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tuberculosis Research Centre, India (Other Government)
Responsible Party: Principal Investigator, Narendran Gopalan, Asst.Director, NIRT, Tuberculosis Research Centre, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRC25
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: HIV Infection; Pulmonary TB
Keywords: TB; HIV; ARR; Short course chemotherapy; Drug resistance
MeSH Terms: conditions — HIV Infections; Tuberculosis, Pulmonary | interventions — Ethambutol; Pyrazinamide; Isoniazid; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2EHRZ3/4HR3 (Active Comparator): Regimen 3. Intermittent - 2EHRZ3/4HR3 (E 1200mg, H 600 mg, R 450/600 mg depending on Weight <60, 600 mg for 60 kg or more, Z 1500 mg given thrice weekly)
  Interventions: Drug: ATT (Ethambutol, Pyrazinamide, INH, Rifampicin)
- 2EHRZ7/4HR7 (Experimental): Regimen 1. Daily - 2EHRZ7/4HR7 (E 800 mg ,H 300 mg, R 450/600 mg depending on Weight <60, 600 mg for 60 kg or more, Z 1500 mg daily)
  Interventions: Drug: ATT (Ethambutol, Pyrazinamide, INH, Rifampicin)
- 2EHRZ7/4HR3 (Experimental): Regimen 2. Part Daily - 2EHRZ7/4HR3 (E 800 mg ,H 300 mg, R 450/600 mg depending on Weight <60, 600 mg for 60 kg or more, Z 1500 mg daily in the intensive phase followed by H-600 mg ,R-450/600 mg in the continuation phase thrice weekly)
  Interventions: Drug: ATT (Ethambutol, Pyrazinamide, INH, Rifampicin)

INTERVENTIONS:
Drug: ATT (Ethambutol, Pyrazinamide, INH, Rifampicin) — Ethambutol 800 mg for daily, 1200 mg for intermittent therapy, Pyrazinamide 1500 mg for both daily and intermittent, INH 300 mg for daily and 600 mg for intermittent therapy, Rifampicin 450 mg for both daily and intermittent therapy for patients below 60 kg, 600 mg for both daily and intermittent therapy for patients 60 kg and above
  Other Names: ATT; Rifampicin

SUMMARY:
Acquired Rifampicin Resistance has emerged as an important issue in the treatment of HIV-TB patients. It has not been a major problem in HIV-negative individuals treated for TB treated with standard intermittent regimens. The study would generate data on the efficacy of daily and thrice weekly regimen of ATT in pulmonary TB patients with HIV in the presence of highly active antiretroviral therapy (HAART). Not many trials have compared sputum conversion and adverse drug reaction between daily and intermittent regimens of ATT in HIV positive patients. This study provides a unique opportunity for comparison of daily and intermittent therapy for HIV patients with pulmonary TB looking into multiple dimensions of HIV-TB treatment namely efficacy, drug resistance, toxicity , drug interaction and immune reconstitution inflammatory syndrome. The primary outcome of the study is to compare the efficacy of three anti-TB regimens in a) reducing bacteriological failures and b) decreasing the emergence of Acquired Rifampicin Resistance (ARR). The secondary outcomes include unfavourable responses (clinical failures, deaths, relapses) as whole, treatment emergent adverse drug reactions, pharmacokinetic levels of ATT and incidence of immune reconstitution syndrome.

DETAILED DESCRIPTION:
HIV positive patients (regardless of ART status) with newly diagnosed pulmonary TB attending the TRC clinics at Chennai, Madurai and Vellore will form the study group. Those who fulfill the clinical inclusion criteria will be evaluated for eligibility to the study after signing a screening consent form. Patients willing to participate in the study will undergo the following investigations namely, sputum examination, chest x-ray, liver and renal function tests. Hematological investigations will include CBC, CD4 and viral load, done periodically at baseline, end of intensive phase of ATT, at the end of TB treatment and once in 6 months during follow-up period of 1 year. Patients getting enrolled in Chennai and its subcentres will also be evaluated for immune reconstitution inflammatory syndrome through additional laboratory investigations. If the patients satisfy the inclusion criteria, a house visit will be done by the social worker to ascertain the facts regarding living condition and domiciliary stability and if continues to remain suitable , will be enrolled into the study after a written, signed and dated informed study consent form. All eligible patients, enrolled into the study, will be randomized to receive one of the three regimens mentioned below. Patients who are ART naïve will be referred to National AIDS Control Organization (NACO) ART centres for assessment and eligibility for procurement of ART according to National guidelines Common opportunistic infections that could occur during study period will be managed according to standard NACO guidelines. Cotrimaxozole DS One tablet once a day will be given to all patients with CD4 < 250 along with multivitamins, unless contraindicated. They will be discharged from the study once their 18th month sputum culture is negative.

Treatment regimens and Dosing:

* Regimen 1. Daily - 2EHRZ7/4HR7 (E 800 mg ,H 300 mg, R 450/600 mg depending on Weight < 60, 600 mg for 60 kg and more, Z 1500 mg daily)
* Regimen 2. Part Daily - 2EHRZ7/4HR3 (E 800 mg ,H 300 mg, R 450/600 mg depending on Weight <60, 600mg for 60 kg and more, Z 1500 mg daily in the intensive phase followed by H-600 mg ,R-450/600 mg in the continuation phase thrice weekly)
* Regimen 3. Intermittent - 2EHRZ3/4HR3 (E 1200mg, H 600 mg, R 450/600 mg depending on Weight < 60, 600 mg for 60 kg and more, Z 1500 mg given thrice weekly)

Statistical design:

Stratification and randomization:

Patients will be stratified based on a) baseline CD4 i) of less than 150 and ii) more than 150 and b) sputum smear grading i) of 0 ,1+ and ii) 2+ , 3+ and randomized to receive one of the three regimens mentioned above, for a period of 6 months, using restricted block scheme. The treatment assignment list will be generated before the start of trial and sequentially numbered sealed opaque envelopes, containing the treatment assigned will be prepared independently in Chennai and Madurai. Assignment of patients to regimens will be done by the study statistician who has no link with the patient.

Sample Size:

Assuming that a daily and a part daily regimen has a 95% resistance- free survival and an intermittent regimen has a 80% resistance free survival during the treatment period, taking into account 20% loss due to death, default and other causes, with a power of 80% and an error of 5%, the sample size was calculated to be 140 per arm (420 cases totally).

Analysis plan Both the efficacy analysis and intent to treat analysis will be undertaken. The primary approach will be intent to treat analysis (ITT) accounting for all patients randomized to study regimen and considering drop outs, deaths and defaulters as unfavourable outcomes. However, Primary MDR -TB will be excluded as an unfavourable response from the ITT analysis despite allocation to study regimen. Efficacy analysis will include only patients who had consumed at least 80 % of the scheduled therapy of ATT. Patients who die within 15 days of starting ATT, and NON-TB deaths during assessment and treatment will not be considered for the efficacy analysis of ATT. Patients who have died during treatment and their cultures grow M.Tb retrospectively will be included as bacteriological failures taking the first event as the outcome. Kaplan Meier survival curves will be constructed and comparison will be done using Log-rank test. To identify the important co-variates in relation to response and toxicity, Cox-regression model will be used. Frailty model will be used to account for individual heterogeneity.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* HIV-1/2 infected patients with Pulmonary TB. This includes sputum smear positive disease.
* Initially smear negative but Xpert-MTB positive or LPA positive taken as a surrogate marker for culture positivity (e.g. miliary TB, Mediastinal adenitis and Chest x-ray with persistent abnormality after antibiotics). as BACTEC (Becton-Dickinson) has been phased out ,Final inclusion will only be patients positive by LJ culture
* Persistent X-ray abnormality will be included for allocation. However final inclusion into both ITT and efficacy analysis will depend on positivity in LJ culture.
* Living within 40 km radius from the nearest sub centre of TRC and willing for attendance as prescribed.
* Likely to remain in the same area for at least one and half years after start of treatment.
* Willing for house visits and surprise checks.
* Willing to participate and give informed consent after going through the terms and conditions of the trial.

Exclusion Criteria:

* Patients with known hypersensitivity to rifampicin
* Pregnancy and lactation at initial presentation
* Major complications like HIV encephalopathy, renal dysfunction (serum creatinine > 1.5 mg% in the absence of dehydration) or jaundice (serum bilirubin > 2 mgs% along with SGOT /SGPT elevation > 2.5 times the upper limit of normal).
* Previous anti-tuberculosis treatment for more than 1 month. Prophylaxis (non-rifampicin containing regimen) will not be considered as prior antituberculosis treatment.
* Moribund, bedridden or unconscious patients.
* Co-morbid conditions like uncontrolled diabetes mellitus, cardiac failure, and malignancy at initial presentation.
* Major psychiatric illness.
* Patients on second line ART, mainly protease inhibitors, at initial presentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2009-09-14 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
unfavourable responses during treatment | At the end of 6 months
  including bacteriological and failures and ARR, clinical failures, TEADRS requiring premanent discontinuation of the drug , Deaths except unnatural and Defaults during treatment period

SECONDARY OUTCOMES:
Unfavorable responses during follow-up | At the end of 6 months and at the end of follow-up of 1 year
  recurrences and deaths during follow up
TEADR's between the groups | At the end of 6 months and at the end of follow-up of 1 year
Incidence of Immune Reconstitution Syndrome among the groups | At the end of 6 months and at the end of follow-up of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Narendran Gopalan, DNB (Chest), Principal Investigator — Scientist 'B', Tuberculosis Research Centre (ICMR), Chennai, India; Soumya Swaminathan, MD, Principal Investigator — Scientist 'F', Tuberculosis Research Centre (ICMR), Chennai, India
Locations (3):
- India (3):
  - Tuberculosis Research Centre (ICMR), Chennai, Tamil Nadu
  - Govt. Hospital of Thoracic Medicine, Tambaram, Chennai, Tamil Nadu
  - Tuberculosis Research Centre (ICMR), Madurai, Tamil Nadu

REFERENCES:
- [Derived] Tiburcio R, Barreto-Duarte B, Naredren G, Queiroz ATL, Anbalagan S, Nayak K, Ravichandran N, Subramani R, Antonelli LRV, Satagopan K, Anbalagan K, Porter BO, Sher A, Swaminathan S, Sereti I, Andrade BB. Dynamics of T-Lymphocyte Activation Related to Paradoxical Tuberculosis-Associated Immune Reconstitution Inflammatory Syndrome in Persons With Advanced HIV. Front Immunol. 2021 Oct 7;12:757843. doi: 10.3389/fimmu.2021.757843. eCollection 2021. PMID 34691079
- [Derived] Gopalan N, Santhanakrishnan RK, Palaniappan AN, Menon PA, Lakshman S, Chandrasekaran P, Sivaramakrishnan GN, Reddy D, Kannabiran BP, Agiboth HKK, Krishnamoorthy V, Rathinam S, Chockalingam C, Manoharan T, Ayyamperumal M, Jayanthi N, Satagopan K, Narayanan R, Krishnaraja R, Sathiyavelu S, Kesavamurthy B, Suresh C, Selvachitiram M, Arasan G, Susaimuthu S, Rathinam P, Angamuthu P, Jayabal L, Murali L, Ramachandran R, Tripathy SP, Swaminathan S. Daily vs Intermittent Antituberculosis Therapy for Pulmonary Tuberculosis in Patients With HIV: A Randomized Clinical Trial. JAMA Intern Med. 2018 Apr 1;178(4):485-493. doi: 10.1001/jamainternmed.2018.0141. PMID 29507938